CLINICAL TRIAL: NCT02566369
Title: A Multi-Center, Randomized, Double-Blind, Parallel-Group Vehicle Controlled Study To Compare The Efficacy And Safety Of CD5789 (Trifarotene) 50μg/g Cream Versus Vehicle Cream In Subjects With Acne Vulgaris
Brief Title: Efficacy and Safety of CD5789 (Trifarotene) 50μg/g Cream Versus Vehicle Cream in Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RD.06.SPR.18251
Record Dates: First submitted 2015-10-01; First posted 2015-10-02 (Estimated); Results first posted 2019-08-22 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2018-07

CONDITIONS: Acne Vulgaris
Keywords: Efficacy; Safety; Acne vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — trifarotene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CD5789 (trifarotene) 50μg/g Cream (Experimental): CD5789 (trifarotene) 50μg/g Cream
  Interventions: Drug: CD5789 (trifarotene) 50μg/g cream
- Placebo Cream (Placebo Comparator): Placebo cream
  Interventions: Drug: Placebo cream

INTERVENTIONS:
Drug: CD5789 (trifarotene) 50μg/g cream — CD5789 (trifarotene) 50µg/g cream applied once daily for 12 weeks.
  Arms: CD5789 (trifarotene) 50μg/g Cream
Drug: Placebo cream — Placebo cream applied once daily for 12 weeks
  Arms: Placebo Cream

SUMMARY:
Assessment of the efficacy and safety of CD5789 (trifarotene) 50μg/g cream applied once daily for 12 weeks in subjects with acne vulgaris.

DETAILED DESCRIPTION:
Clinical Trial for each subject is approximately 14 weeks and are randomized to one of the two treatments for 12 weeks. Subjects must be 9 years of age and older with acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* The subject is a male or female, 9 years of age or older, at Screening visit.
* The Subject has moderate acne at Screening and Baseline.
* The subject is a female of non childbearing potential
* The subject is a female of childbearing potential with a negative pregnancy test and who is strictly abstinent or who agrees to use an effective and approved contraceptive method for the duration of the study and at least 1 month after the last study drug application.

Exclusion Criteria:

* The subject has severe forms of acne (e.g., acne conglobate, acne fulminant) or secondary acne form (e.g.,chloracne, drug-induced acne, etc.).
* The subject has any uncontrolled or serious disease or any medical or surgical condition that may either interfere with the interpretation of the trial results and/or put the subject at significant risk (according to the Investigator's judgment) if the subject takes part to the trial.
* The subject has been exposed to excessive ultraviolet (UV) radiation within one month prior to the Baseline visit or the subject is planning intense UV exposure during the study (i.e., occupational exposure to the sun, sunbathing, tanning salon use, phototherapy, etc.)
* The subject is unwilling to refrain from use of prohibited medication during the clinical trial

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1208 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2017-11-14 (Actual); Study Completion 2017-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Tan, MD, Principal Investigator — Windsor Clinical Research; Ulrike Blume-Peytavi, MD, Principal Investigator — Charité Universitätsmedizin
Locations (124):
- United States (86):
  - Galderma Investigational Site (8258), Mobile, Alabama
  - Galderma Investigational Site (# 8530), Glendale, Arizona
  - Galderma Investigational Site (# 8511), Phoenix, Arizona
  - Galderma Investigational Site (# 8009), Hot Springs, Arkansas
  - Galderma Investigational Site (# 8355), Rogers, Arkansas
  - Galderma Investigational Site (# 8456), Beverly Hills, California
  - Galderma Investigational site (8578), Cerritos, California
  - Galderma Investigational Site (# 8526), Clovis, California
  - Galderma Investigational Site (8577), Encinitas, California
  - Galderma Investigational Site (# 8224), Fremont, California
  - Galderma Investigational Site (# 8509), Fullerton, California
  - Galderma Investigational Site (# 8507), Huntington Beach, California
  - Galderma Investigational Site (# 8425), Newport Beach, California
  - Galderma Investigational Site (# 8052), Oceanside, California
  - Galderma Investigational Site (# 8528), Santa Ana, California
  - Galderma Investigational Site (# 8160), Santa Monica, California
  - Galderma Investigational Site (# 8443), Temecula, California
  - Galderma Investigational Site (8572), Colorado Springs, Colorado
  - Galderma Investigational Site (# 8510), Englewood, Colorado
  - Galderma Investigational Site (# 8370), Boynton Beach, Florida
  - Galderma Investigational Site (# 8543), Fort Lauderdale, Florida
  - Galderma Investigational Site (8143), Miami, Florida
  - Galderma Investigational site (8259), Miramar, Florida
  - Galderma Investigational Site (# 8522), North Miami Beach, Florida
  - Galderma Investigational Site (# 8531), Orange Park, Florida
  - Galderma Investigational Site (8502), Orlando, Florida
  - Galderma Investigational Site (#8213), Ormond Beach, Florida
  - Galderma Investigational Site (# 8529), Sanford, Florida
  - Galderma Investigational Site (# 8455), St. Petersburg, Florida
  - Galderma Investigational Site (# 8523), Tampa, Florida
  - Galderma Investigational Site (# 8126), West Palm Beach, Florida
  - Galderma Investigational Site (#8189), Snellville, Georgia
  - Galderma Investigational Site (8582), Idaho Falls, Idaho
  - Galderma Investigational Site (# 8367), Arlington Heights, Illinois
  - Galderma Investigational Site (8191), Chicago, Illinois
  - Galderma Investigational site (8571), Darien, Illinois
  - Galderma Investigational Site (8575), Oakbrook Terrace, Illinois
  - Galderma Investigational Site (# 8366), Plainfield, Indiana
  - Galderma Investigational Site (# 8532), Overland Park, Kansas
  - Galderma Investigational Site (# 8069), Louisville, Kentucky
  - Galderma Investigational Site (8092), Louisville, Kentucky
  - Galderma Investigational Site (8545), Owensboro, Kentucky
  - Galderma Investigational Site (8457), Monroe, Louisiana
  - Galderma Investigational site (8580), New Orleans, Louisiana
  - Galderma Investigational Site (# 8012), Glenn Dale, Maryland
  - Galderma Investigational Site (# 8525), Rockville, Maryland
  - Galderma Investigational Site (# 8541), Quincy, Massachusetts
  - Galderma Investigational Site (#8512), Bay City, Michigan
  - Galderma Investigational Site (8574), Clarkston, Michigan
  - Galderma Investigational Site (#8033), Clinton Township, Michigan
  - Galderma Investigational Site (8129), Fort Gratiot, Michigan
  - Galderma Investigational Site (# 8226), Warren, Michigan
  - Galderma Investigational Site (# 8521), Saint Joseph, Missouri
  - Galderma Investigational Site (#8027), St Louis, Missouri
  - Galderma Investigational Site (# 8544), Lincoln, Nebraska
  - Galderma Investigational Site (# 8108), Las Vegas, Nevada
  - Galderma Investigational Site (#8420), Newington, New Hampshire
  - Galderma Investigational Site (# 8506), Hackensack, New Jersey
  - Galderma Investigational Site (#8500), Brooklyn, New York
  - Galderma Investigational Site (8524), East Setauket, New York
  - Galderma Investigational Site (8568), New York, New York
  - Galderma Investigational Site (8585), New York, New York
  - Galderma Investigational Site (8279), New York, New York
  - Galderma Investigational Site (8566), Charlotte, North Carolina
  - Galderma Investigational Site (#8514), Hickory, North Carolina
  - Galderma Investigational Site (# 8195), Beachwood, Ohio
  - Galderma Investigational Site (# 8016), Cincinnati, Ohio
  - Galderma Investigational site (8595), Dublin, Ohio
  - Galderma Investigational Site (8188), Hershey, Pennsylvania
  - Galderma Investigational site (8353), Yardley, Pennsylvania
  - Galderma Investigational Site (# 8369), Charleston, South Carolina
  - Galderma Investigational Site (# 8117), Knoxville, Tennessee
  - Galderma Investigational Site (# 8515), Nashville, Tennessee
  - Galderma Investigational Site (# 8542), Arlington, Texas
  - Galderma Investigational Site (#8513), Austin, Texas
  - Galderma Investigational site (8579), Beaumont, Texas
  - Galderma Investigational Site (# 8245), Dallas, Texas
  - Galderma Investigational Site (8183), Houston, Texas
  - Galderma Investigational site (8576), Katy, Texas
  - Galderma Investigational Site (8583), Murphy, Texas
  - Galderma Investigational Site (8567), San Antonio, Texas
  - Galderma Investigational site (8433), San Antonio, Texas
  - Galderma Investigational site (8329), San Antonio, Texas
  - Galderma Investigational site (8106), Layton, Utah
  - Galderma Investigational Site (# 8214), Salt Lake City, Utah
  - Galderma Investigational Site (# 8351), Seattle, Washington
- Canada (13):
  - Galderma Investigational Site (# 8215), Calgary, Alberta
  - Galderma Investigational site (8161), Surrey, British Columbia
  - Galderma Investigational Site (# 8154), Winnipeg, Manitoba
  - Galderma Investigational Site (8586), Barrie, Ontario
  - Galderma Investigational Site (# 8038), Hamilton, Ontario
  - Galderma Investigational Site (# 8426), London, Ontario
  - Galderma Investigational Site (# 8026), Markham, Ontario
  - Galderma Investigational Site (# 8135), North Bay, Ontario
  - Galderma Investigational Site (# 8168), Oakville, Ontario
  - Galderma Investigational Site (# 8340), Peterborough, Ontario
  - Galderma Investigational Site (# 8338), Richmond Hill, Ontario
  - Galderma Investigational Site (8001), Waterloo, Ontario
  - Galderma Investigational Site (# 8060), Windsor, Ontario
- Germany (12):
  - Galderma Investigational Site (5566), Augsburg
  - Galderma Investigational Site (5604), Berlin
  - Galderma Investigational Site (5815), Berlin
  - Galderma Investigational Site (5750), Darmstadt
  - Galderma Investigational Site (5572), Dessau
  - Galderma Investigational Site (5204), Dresden
  - Galderma Investigational Site (5434), Dresden
  - Galderma Investigational Site (5146), Eberstadt
  - Galderma Investigational Site (5838), Hamburg
  - Galderma Investigational Site (5635), Langenau
  - Galderma Investigational Site (5543), Mainz
  - Galderma Investigational Site (5307), Münster
- Hungary (9):
  - Galderma Investigational Site (5802), Balatonfüred
  - Galderma Investigational Site (5567), Budapest
  - Galderma Investigational Site (5812), Budapest
  - Galderma Investigational Site (5685), Cegléd
  - Galderma Investigational Site (5254), Nyíregyháza
  - Galderma Investigational Site (5811), Pécel
  - Galderma Investigational Site (5263), Püspökladány
  - Galderma Investigational Site (5237), Szeged
  - Galderma Investigational Site (5767), Szekszàrd
- Puerto Rico (4):
  - Galderma Investigational Site (8592), Aibonito
  - Galderma Investigational Site (8594), Caguas
  - Galderma Investigational site (8100), Carolina
  - Galderma Investigational Site (8593), San Juan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CD5789 (Trifarotene) 50μg/g Cream | Placebo Cream
Started | 612 | 596
Completed | 540 | 535
Not Completed | 72 | 61

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CD5789 (Trifarotene) 50μg/g Cream | Placebo Cream | Total
Number analyzed (Participants) | 612 | 596 | 1208
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 314 | 278 | 592
  Between 18 and 65 years | 298 | 318 | 616
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 305 | 324 | 629
  Male | 307 | 272 | 579
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 135 | 148 | 283
  Not Hispanic or Latino | 477 | 448 | 925
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11 | 5 | 16
  Asian | 23 | 32 | 55
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 47 | 49 | 96
  White | 508 | 484 | 992
  More than one race | 8 | 10 | 18
  Unknown or Not Reported | 14 | 15 | 29
Region of Enrollment [Number; unit: participants]
  Canada | 70 | 69 | 139
  Puerto Rico | 27 | 28 | 55
  Hungary | 44 | 44 | 88
  United States | 407 | 395 | 802
  Germany | 64 | 60 | 124
Physician Global Assessment Scale Face [Count of Participants; unit: Participants] — 0 - Clear (Clear skin with no inflammatory or non-inflammatory lesions.)
  1. - Almost Clear (A few scattered comedones and a few small papules.)
  2. - Mild (Easily recognizable; less than half the surface is involved. Some comedones and some papules and pustules.)
  3. - Moderate (More than half of the surface is involved. Many comedones, papules and pustules. One nodule may be present.)
  4. - Severe (Entire surface is involved. Covered with comedones, numerous papules and pustules. Few nodules may be present.)
  Participants
    Clear | 0 | 0 | 0
    Almost Clear | 0 | 0 | 0
    Mild | 0 | 0 | 0
    Moderate | 612 | 596 | 1208
    Severe | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Investigator Global Assessment (IGA) Success Rate at Week 12
Description: Number of subjects who achieved an Investigator Global Assessment (IGA) score of 1 (almost clear) or 0 (Clear) and at least a 2-grade improvement from Baseline to Week 12.
Time Frame: From Baseline to Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | CD5789 (Trifarotene) 50μg/g Cream | Placebo Cream
Number analyzed (Participants) | 612 | 596
Participants | 180 | 116

ADVERSE EVENTS:
Time Frame: Each participant's adverse events were collected starting at the first visit (screening) until the last visit (Week 12).
Arm/Group | CD5789 (Trifarotene) 50μg/g Cream | Placebo Cream
All-Cause Mortality (participants affected / at risk) | 0/612 | 0/596
Serious Adverse Events (participants affected / at risk) | 4/612 | 2/596
Other Adverse Events (participants affected / at risk) | 177/612 | 74/596
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CD5789 (Trifarotene) 50μg/g Cream (N=612) | Placebo Cream (N=596)
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hereditary angioedema (Congenital, familial and genetic disorders) | 0 | 1
Procedural dizziness (Injury, poisoning and procedural complications) | 1 | 0
Urinary Tract Infection (Renal and urinary disorders) | 0 | 1
Infectious Mononucleosis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Atypical Pneumonia (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CD5789 (Trifarotene) 50μg/g Cream (N=612) | Placebo Cream (N=596)
Sunburn (Injury, poisoning and procedural complications) | 27 | 5
Headache (Nervous system disorders) | 6 | 12
Application Site Irritation (General disorders) | 66 | 4
Application Site Pruritis (General disorders) | 24 | 8
Skin Irritation (Skin and subcutaneous tissue disorders) | 8 | 0
Nasopharyngitis (Infections and infestations) | 24 | 27
Upper Respiratory Tract Infection (Infections and infestations) | 10 | 8
Influenza (Infections and infestations) | 6 | 9
Sinusitis (Infections and infestations) | 6 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-03-10): https://cdn.clinicaltrials.gov/large-docs/69/NCT02566369/Prot_000.pdf
  • Statistical Analysis Plan (2015-10-05): https://cdn.clinicaltrials.gov/large-docs/69/NCT02566369/SAP_002.pdf